CLINICAL TRIAL: NCT06874296
Title: Pilot, Open, Prospective, Randomized, Multicenter Trial On Quality Assessment Of Declined Liver Grafts By Normothermic Ex Vivo Machine Perfusion For Decreasing Time To Transplantation
Brief Title: Assessing Declined Liver Grafts With Normothermic Machine Perfusion to Reduce Transplant Waiting Time
Acronym: ExTra
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Nathanael Raschzok, Principal Investigator, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20024292; 543051616 (Other: German Research Foundation)
Record Dates: First submitted 2025-02-27; First posted 2025-03-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Liver Transplantation; Liver Diseases; Surgery
Keywords: Liver Transplantation; Extended Criteria Donors; Normothermic Machine Perfusion; Discarded Liver Grafts
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: The treatment in the intervention arm will be available for patient for 12 months after randomization. Patients who have not yet received a graft after 12 months and are therefore still on the waiting list are administratively censored.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (No Intervention): Patient will be listed for liver transplantation through standard allocation only.
- ExTra Option (Experimental): Patients will receive the option to receive a graft that was declined by all German Transplant Centers but meets predefined quality criteria during at least 4 hours of normothermic machine perfusion (ExTra-LT) or a liver via regular allocation - whichever occurs first.
  Declined liver grafts will be allocated based on Eurotransplant's first-come-first-serve principle, with consideration for transport logistics and recipient eligibility. Only grafts meeting the following criteria will be considered: Macrovesicular steatosis <60%, fibrosis grade ≤F3, no histopathologic evidence of cirrhosis, graft weight between 1-2.5 kg, no previous machine perfusion preservation.
  Interventions: Device: Quality Assessment with Normothermic Machine Perfusion (NMP)

INTERVENTIONS:
Device: Quality Assessment with Normothermic Machine Perfusion (NMP) — Quality assessment using NMP in the experimental arm is performed according to previously published viability criteria for initially declined liver grafts, which are mandatory for all participating study centers, with minor device-specific modifications. These criteria are based on the Birmingham criteria used in the VITTAL trial for viability assessment of DBD and DCD grafts with the OrganOx Metra device and are comparable to the Groningen criteria used with the LiverAssist and PerLife device, with the exception of biliary viability.
  These criteria are: Lactate clearance < 2.5 mmol/L, And two or more of the following: Evidence of bile production, maintenance of a perfusate pH >7.30 (without correction for at least one hour), glucose metabolism (falling perfusate glucose value with consistent downward trend), maintenance of stable arterial and portal venous flows (OrganOx Metra: 150 and 500 mL/min respectively), homogeneous perfusion with soft consistency of the parenchyma.
  Arms: ExTra Option

SUMMARY:
The goal of this study is to find out if quality assessment by normothermic machine perfusion can be used to safely increase the number of usable donor livers, helping more people get transplants faster and with better results. This process keeps a donated liver working outside the body before transplantation, allowing surgeons to assess whether livers previously considered unsuitable can still be used.

The main questions this study aims to answer are:

* Does this method help patients get a transplant sooner?
* Can this method make more livers available for transplant?
* Does it improve survival and health after transplant?

Participants in this study must be on the waiting list for a liver transplant with a ReMELD-Na-Score of 21 or less (equivalent to MELD ≤25) and must not qualify for certain special exceptions. Participants will be randomly placed into one of two groups:

* Experimental group: In addition to regular organ offers, these participants may receive a liver that was initially not considered for transplantation but meets quality standards after at least four hours of machine perfusion.
* Control group: These participants will receive a liver through the usual transplant process.

The main measure of success is how quickly participants receive a transplant. Researchers will also look at other important factors, such as survival rates, quality of life, hospital stay, and complications after transplant.

This study may help improve liver transplantation by making better use of available donor livers, reducing waiting times, and improving patient outcomes.

DETAILED DESCRIPTION:
Liver transplantation is the treatment of choice for patients with advanced liver cirrhosis, hepatocellular carcinoma within the Milan criteria, and severe metabolic or autoimmune liver diseases. However, organ shortage remains a significant issue, particularly in Germany, where only 58% of patients on the waiting list received a transplant in 2022. Patients with MELD ≤25, who are ineligible for [Non]-Standard Exception criteria, face particularly long waiting times and lower transplant rates.

Despite the shortage, approximately 24% of all liver grafts in Germany are declined due to donor age, macrosteatosis, or prolonged cold ischemia. Emerging technologies, such as NMP, allow for objective graft quality assessment before transplantation. Several non-randomized studies in the UK, Netherlands, Australia, and the USA have demonstrated the potential of NMP to increase organ utilization. The ExTra trial is the first randomized controlled study to investigate whether declined liver grafts, following NMP-based quality assessment, can safely and effectively reduce the waiting time for patients with ReMELD-Na-Score ≤ 21(equivalent to MELD ≤25).

ELIGIBILITY:
Inclusion Criteria:

* Able to consent
* ≥ 18 years old
* Listed in status "transplantable" by the transplant conference of the study centre for liver transplantation, according to the guidelines of the German Medical Association valid at the time of inclusion
* ReMELD-Na-Score ≤ 21 (equivalent to MELD ≤25), not eligible for [non]standard exceptions
* Medically suitable and informed for transplantation with an organ that fulfils extended donor criteria (Eurotransplant ECD criteria)
* Patient information and written consent to participate in the Extra trial
* No participation in another interventional study during participation

Exclusion Criteria:

* Listed for retransplantation
* High-Urgency Listing
* Listed for combined organ transplantation
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Time-to-Transplant | From date of randomization to liver transplantation (up to 12 months after date of randomization)

SECONDARY OUTCOMES:
Death | From date of randomization to death (up to 12 months after date of randomization)
  Patient death during the 12-month intervention period, regardless of liver transplantation or not.
Disease Progression | From date of randomization to event (up to 12 months after date of randomization)
  Change of ReMELD-Na-Score above 21 while listed as "transplantable" on the waitlist. Occurence of new contraindication for liver transplantation
Proportion of Patients Recovered on the Waitlist | From date of randomization to event (up to 12 months after date of randomization)
  Proportion of patients with change in overall health that no liver transplantation is further required in relation to all patients on the waitlist in the trial.
Number of patients listed for transplantation after 12 months | 12 months after randomization
  Number of patients listed for transplantation after 12 months.
Overall patient survival | From date of randomization to death (up to 24 months after date of randomization)
  Overall patient survival in the study.
Patient-reported Quality of Life | up to 24 months
  Patient-reported Quality of Life measured in the EuroQOL EQ5DL. Two aspects will be reported: The EuroQOL visual analog scale (EQ VAS) on a scale from 0-100 points and the proportion of responses by level of severity for the five EQ-5D-5L dimensions (each reported on a five level scale).
Graft utilization rate | up to 12 months
  Proportion of used livers of all organs offered to patients on the waiting list
Inpatient Costs for Liver Transplantation | First 90 days after liver transplantation
  Analysis of liver transplantation-associated costs. This will be total costs, earnings and profit measured in Euros (EUR) for the primary inpatient stay of liver transplantation.

OTHER OUTCOMES:
3-month Graft Survival | Within 3 months after date of liver transplantation
  Graft survival is defined as the need for retransplantation within the first 3 months after liver transplantation. This is one of the "Safety" endpoints and will be evaluated by the Data Safety Monitoring Board.
3-month Patient Survival | Within 3 months after date of liver transplantation
  Patient survival is defined as death within the first 3 months after liver transplantation. This is one of the "Safety" endpoints and will be evaluated by the Data Safety Monitoring Board.
Patient Survival | 12 months after liver transplantation
  Patient Survival after liver transplantation
Early graft function | Until 10 days after liver transplantation
  Early graft function measured by the Early Allograft Failure Simplified Estimation (EASE) Score on a scale from -6 (extremely low risk) to +6 (unsustainable risk).
Intensive Care Unit Stay | First 30 days after liver transplantation
  Length of stay on the intensive care unit in days.
Length of Hospital Stay | First 90 days after liver transplantation
  Total duration of days spent in the hospital after liver transplantation.
Comprehensive Complication Index | Until 90 days after liver transplantation
  Post-transplant Comprehensive Complication Index, measured on a scale of 0-100, to quantify procedure related morbidity.
Biliary Complications | Until 12 months after liver transplantation
  Ischemic-Type Biliary Lesions (clinically and as part of the planned MRCP 12 months after liver transplantation)
Graft Survival | 12 months after liver transplantation
  Graft survival after liver transplantation.
Acceptance Rate | Until 12 months after randomization
  1 / number of unrealized organ offers [accepted for the patient either primarily or within the extended/rescue allocation but not transplanted]
Graft-Rescue Rate | Until 12 months after randomization
  Livers that meet quality criteria during NMP / all organs assessed through NMP in the study
Risk of Graft Loss | On day of liver transplantation (within the 12 month intervention period after date of randomization)
  Risk of early graft loss as measured by the Balance of Risk (BAR) Score on a scale from 0-27.

CONTACTS AND LOCATIONS:
Locations (9):
- Germany (9):
  - University Medical Center Hamburg-Eppendorf, Hamburg, Hamburg
  - University Hospital RWTH Aachen, Aachen, North Rhine-Westphalia
  - University Hospital Bonn, Bonn, North Rhine-Westphalia
  - University Hospital Muenster, Münster, North Rhine-Westphalia
  - Department of Surgery Campus Charité Mitte | Campus Virchow-Klinikum, Charité - Universitätsmedizin Berlin, Berlin, State of Berlin
  - Department of General, Visceral and Transplantation Surgery, LMU University Hospital, LMU Munich, München
  - Department of Surgery, University Hospital Regensburg, Regensburg
  - Eberhard Karls University of Tübingen, Department of General Visceral and Transplant Surgery, Tübingen
  - Department of General, Visceral, Transplantation, Vascular, and Pediatric Surgery, University Hospital Wurzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared due to data protection regulations and ethical considerations. Given the sensitive nature of the data, strict confidentiality measures must be maintained to protect participants' privacy. Compliance with GDPR and institutional policies prevents the disclosure of personally identifiable information, ensuring that data handling aligns with legal and ethical standards.

REFERENCES:
- See also: Official Trial Homepage — https://extra-trial.de/en_home/
- See also: Funding Information — https://gepris.dfg.de/gepris/projekt/543051616